CLINICAL TRIAL: NCT01494922
Title: A PHASE 2, OPEN-LABEL STUDY TO PROVIDE REVISION OF SCARS RESULTING FROM SURGERY IN PRIOR STUDIES OF EXC 001
Brief Title: Safety and Efficacy of EXC 001 in Subjects Who Have Participated in Prior Studies of EXC 001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EXC 001-206; B5301003 (Other: Alias Study Number)
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Results first posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Reduction in Severity of Skin Scarring
Keywords: Skin scarring; cicatrix; hypertrophic scar; hypertrophic scar prevention
MeSH Terms: conditions — Cicatrix; Cicatrix, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label (Experimental)
  Interventions: Drug: EXC 001 (currently called PF-06473871)

INTERVENTIONS:
Drug: EXC 001 (currently called PF-06473871) — Single dose administered by injection at four different times

SUMMARY:
The purpose of this study is to provide subjects who participated in prior studies of EXC 001 the opportunity to have their hypertrophic scars surgically revised and treated with EXC 001.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults who have participated in previous studies of EXC 001.
* Healthy adults who have chosen to have their scars revised.

Exclusion Criteria:

* Currently pregnant or pregnant during the 6 months prior to inclusion in the study, or breast feeding.
* Participation in another clinical trial within 30 days prior to the start of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-12-08 (Actual); Primary Completion 2013-09-10 (Actual); Study Completion 2013-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Altus Research, Lake Worth, Florida
  - Northwestern University,Division of Plastic Surgery, Chicago, Illinois
  - Jewell Plastic Surgery Center, Eugene, Oregon
  - Connall Consmetic Surgery, Tualatin, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=EXC001-206&StudyName=Safety%20and%20Efficacy%20of%20EXC%20001%20in%20Subjects%20Who%20Have%20Participated%20in%20Prior%20Studies%20of%20EXC%20001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who participated in any of the previous studies (EXC 001-202 [NCT01037985], EXC 001-203 [NCT01037413] and EXC 001-204 [NCT01346969]), had scars at a minimum of 1 year after surgery in previous study which qualified for scar revision and chose scar revision treatment with EXC 001 (PF-06473871) were eligible for this study.
Groups:
- EXC 001 (PF-06473871): Participants who underwent scar revision surgery on Day 1 and received 4 intradermal injections of EXC 001 (PF-06473871) at a dose of 5 milligram per centimeter (mg/cm) at Week 2, 5, 8 and 11 after the surgical incision was closed, to both sides of the incision/scar. Participants received treatment for total scar length of up to 14 centimeter (cm).
Period: Overall Study
Arm/Group | EXC 001 (PF-06473871)
Started | 14
Completed | 13
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who completed the scar revision surgery (Day 1 visit).
Groups:
- EXC 001 (PF-06473871): Participants who underwent scar revision surgery on Day 1 and received 4 intradermal injections of EXC 001 (PF-06473871) at a dose of 5 mg/cm at Week 2, 5, 8 and 11 after the surgical incision was closed, to both sides of the incision/scar. Participants received treatment for total scar length of up to 14 cm.
Arm/Group | EXC 001 (PF-06473871)
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (7.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included SAEs and all non-SAEs that occurred during the study.
Time Frame: Week 2 to Week 24
Population: Safety population included all participants who completed the scar revision surgery (Day 1 visit).
Measure: Count of Participants; unit: Participants
Arm/Group | EXC 001 (PF-06473871)
Number analyzed (Participants) | 14
Participants
  AEs | 8
  SAEs | 0

2. Primary Outcome: Number of Participants With Positive Skin Sensitivity Reaction
Description: Participants were instructed to inform the investigator in case of any itching, redness, pain or any other symptom that appeared to be a rash at the injection sites. Erythematous, raised (indurated) and edematous reactions were considered as positive skin sensitivity reactions. In this outcome measure number of participants with any positive skin sensitivity reaction were reported.
Time Frame: Day 1 up to Week 24
Population: Safety population included all participants who completed the scar revision surgery (Day 1 visit).
Measure: Count of Participants; unit: Participants
Arm/Group | EXC 001 (PF-06473871)
Number analyzed (Participants) | 14
Participants | 2

3. Primary Outcome: Number of Participants With Clinically Significant Findings in Laboratory Examinations
Description: Following parameters were analyzed for laboratory examination: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); Hepatobiliary biochemistry: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Albumin, Alkaline Phosphatase, Total Bilirubin ; Renal Function Tests: Blood Urea Nitrogen (BUN), Creatinine, Creatinine Kinase, Uric Acid ; Electrolytes: Sodium, Potassium; Glucose; Urine analysis: (decimal logarithm of reciprocal of hydrogen ion activity )[pH], Specific gravity. Clinically significant laboratory abnormality findings were based on investigator discretion.
Time Frame: Day 1 up to Week 24
Population: Safety population included all participants who completed the scar revision surgery (Day 1 visit).
Measure: Count of Participants; unit: Participants
Arm/Group | EXC 001 (PF-06473871)
Number analyzed (Participants) | 14
Participants | 0

4. Primary Outcome: Number of Participants With Clinically Significant Change in Vital Signs
Description: Following vital sign parameters were assessed: diastolic blood pressure, systolic blood pressure, respiration rate, pulse rate, temperature and body weight. Number of participants with clinically significant change in any vital sign parameter compared to baseline were reported. Clinically significant change in vital signs criteria were based on investigator's discretion.
Time Frame: Day 1 up to Week 24
Population: Safety population included all participants who completed the scar revision surgery (Day 1 visit).
Measure: Count of Participants; unit: Participants
Arm/Group | EXC 001 (PF-06473871)
Number analyzed (Participants) | 14
Participants | 0

5. Primary Outcome: Number of Participants With Clinically Significant Findings in Electrocardiogram (ECG) Abnormalities
Description: Following parameters were analyzed: heart rate, PR interval, QT interval, QRS interval and QT interval corrected using Fridericia's formula (QTcF). Clinically significant findings in ECG were based on investigator's discretion.
Time Frame: Day 1 up to Week 24
Population: Safety population included all participants who completed the scar revision surgery (Day 1 visit).
Measure: Count of Participants; unit: Participants
Arm/Group | EXC 001 (PF-06473871)
Number analyzed (Participants) | 14
Participants | 0

6. Primary Outcome: Number of Participants With Abnormalities in Physical Examinations
Description: Physical examination included the assessment of skin, head, ears, eyes, nose, throat, respiratory system, cardiovascular system, abdomen (including liver and kidneys), musculoskeletal system, neurological system, gastrointestinal system, genitourinary system, endocrine system and lymph nodes. Abnormality in physical examination were based on investigator's discretion.
Time Frame: Day 1 up to Week 24
Population: Safety population included all participants who completed the scar revision surgery (Day 1 visit).
Measure: Count of Participants; unit: Participants
Arm/Group | EXC 001 (PF-06473871)
Number analyzed (Participants) | 14
Participants | 3

7. Secondary Outcome: Physician Observer Scar Assessment Score: Individual Sub Scores and Composite Score
Description: Physician assessment of scar was done using a valid published 10-point rating scale. Assessment included following sub scores: vascularity, pigmentation, thickness, relief, pliability, surface area and overall opinion for scar, on a score of 1 = normal skin to 10 = worst scar imaginable. Composite score was the sum of all the sub scores except the overall opinion score and range from 6 (best score) to 60 (worst score).
Time Frame: Week 24
Population: Analysis population included all participants who completed Week 24 efficacy assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EXC 001 (PF-06473871)
Number analyzed (Participants) | 13
units on a scale
  Overall opinion | 4.63 (2.033)
  Vascularity | 4.02 (1.838)
  Pigmentation | 3.83 (1.848)
  Thickness | 4.55 (2.022)
  Relief | 4.06 (2.112)
  Pliability | 3.97 (1.932)
  Surface area | 4.71 (1.534)
  Composite Score | 25.15 (8.744)

8. Secondary Outcome: Participant Observer Scar Assessment Score: Individual Sub Scores, Composite Score, Scar Appearance Composite Score
Description: Participants rated pain, itching, color, stiffness, thickness, irregularity and overall opinion of scar on 10-point scale. For pain and itching associated with scar: range = 1 (no, not at all) to 10 (yes, worst imaginable) and for other parameters associated with scar compared to normal skin: range = 1 (no, same as normal skin) to 10 (yes, very different). Composite score is the sum of all sub scores except overall opinion, range 6 (best) to 60 (worst). Scar appearance composite score is the sum of all sub scores except overall opinion, pain and itching, range 4 (best) to 40 (worst).
Time Frame: Week 24
Population: Analysis population included all participants who completed Week 24 efficacy assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EXC 001 (PF-06473871)
Number analyzed (Participants) | 13
units on a scale
  Overall opinion | 6.21 (2.660)
  Pain | 2.46 (1.620)
  Itching | 2.03 (1.234)
  Color | 6.72 (2.323)
  Stiffness | 5.76 (2.487)
  Thickness | 5.56 (2.508)
  Irregular | 5.62 (2.494)
  Composite Score | 28.15 (10.457)
  Scar Appearance composite Score | 23.67 (9.110)

9. Secondary Outcome: Number of Scars Classified According to Physician Photonumeric Guide Score Severity Category
Description: Physician rated severity of each scar using a photonumeric guide on a scale range from 1 to 5 (where 1 = minimal, 2 = mild, 3 = moderate, 4 = severe, 5 = very severe). Number of scars with different ratings of scar severity were reported. Participants may have received treatment for multiple scars (up to 5 scars), results are reported for all scars (individual scar) and most severe scar for all the participants.
Time Frame: Week 24
Population: Analysis population included all participants who completed Week 24 efficacy assessments. Here, "type of unit analyzed" signifies number of scars evaluable.
Measure: Number; unit: scars
Units Other Than Participants: scars
Arm/Group | EXC 001 (PF-06473871)
Number analyzed (Participants) | 13
Number analyzed (scars) | 28
scars
  Individual Scar: Minimal | 5
  Individual Scar: Mild | 12
  Individual Scar: Moderate | 4
  Individual Scar: Severe | 1
  Individual Scar: Very Severe | 6
  Most Severe Scar: Minimal: number analyzed (scars) | 13
  Most Severe Scar: Minimal | 2
  Most Severe Scar: Mild: number analyzed (scars) | 13
  Most Severe Scar: Mild | 4
  Most Severe Scar: Moderate: number analyzed (scars) | 13
  Most Severe Scar: Moderate | 2
  Most Severe Scar: Severe: number analyzed (scars) | 13
  Most Severe Scar: Severe | 1
  Most Severe Scar: Very Severe: number analyzed (scars) | 13
  Most Severe Scar: Very Severe | 4

10. Secondary Outcome: Number of Scars Classified According to Subject Participant Photonumeric Guide Score Severity Category
Description: Participants rated severity of each scar using a photonumeric guide on a scale range from 1 to 5 (where 1 = minimal, 2 = mild, 3 = moderate, 4 = severe, 5 = very severe). Number of scars with different ratings of scar severity were reported. Participants may have received treatment for multiple scars (up to 5 scars), results are reported for all scars (individual scar) and most severe scar for all the participants.
Time Frame: Week 24
Population: as for outcome 9
Measure: Number; unit: scars
Units Other Than Participants: scars
Arm/Group | EXC 001 (PF-06473871)
Number analyzed (Participants) | 13
Number analyzed (scars) | 28
scars
  Individual Scar: Minimal | 6
  Individual Scar: Mild | 7
  Individual Scar: Moderate | 6
  Individual Scar: Severe | 3
  Individual Scar: Very Severe | 6
  Most Severe Scar: Minimal: number analyzed (scars) | 13
  Most Severe Scar: Minimal | 2
  Most Severe Scar: Mild: number analyzed (scars) | 13
  Most Severe Scar: Mild | 1
  Most Severe Scar: Moderate: number analyzed (scars) | 13
  Most Severe Scar: Moderate | 4
  Most Severe Scar: Severe: number analyzed (scars) | 13
  Most Severe Scar: Severe | 1
  Most Severe Scar: Very Severe: number analyzed (scars) | 13
  Most Severe Scar: Very Severe | 5

ADVERSE EVENTS:
Time Frame: Week 2 to Week 24
Arm/Group | EXC 001 (PF-06473871)
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 8/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EXC 001 (PF-06473871) (N=14)
Sinusitis (Infections and infestations) | 1
Fungal Infection (Infections and infestations) | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Injection site erythema (General disorders) | 2
Injection site induration (General disorders) | 1
Injection site pain (General disorders) | 1
Injection site pruritus (General disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Lip swelling (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Headache (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.